CLINICAL TRIAL: NCT00392834
Title: Prospective Phase II Study of a High Dose, Short Course Regimen (R-CODOX-M/IVAC) Including CNS Penetration and Intensive IT Prophylaxis in HIV-Associated Burkitt's and Atypical Burkitt's Lymphoma
Brief Title: Rituximab and Combination Chemotherapy in Treating Patients With Newly Diagnosed, HIV-Associated Burkitt's Lymphoma
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: AIDS Malignancy Consortium (Network)
Collaborators: National Cancer Institute (NCI) (NIH); The Emmes Company, LLC (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: AMC-048; U01CA070019 (NIH); CDR0000510918 (Other: NCI)
Record Dates: First submitted 2006-10-25; First posted 2006-10-26 (Estimated); Results first posted 2013-02-28 (Estimated); Last update posted 2018-06-06 (Actual); Status verified 2018-05

CONDITIONS: Lymphoma
Keywords: stage I adult Burkitt lymphoma; stage III adult Burkitt lymphoma; stage IV adult Burkitt lymphoma; contiguous stage II adult Burkitt lymphoma; noncontiguous stage II adult Burkitt lymphoma; AIDS-related peripheral/systemic lymphoma
MeSH Terms: conditions — Lymphoma; Burkitt Lymphoma | interventions — Filgrastim; pegfilgrastim; Rituximab; Cyclophosphamide; Cytarabine; Doxorubicin; Etoposide; Ifosfamide; Leucovorin; Methotrexate; Hydrocortisone; Vincristine

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Regimen A (R-CODOX-M chemotherapy) (Experimental): Patients receive rituximab IV and doxorubicin hydrochloride IV over 15 minutes on day 1, cyclophosphamide IV over 30-60 minutes on days 1 and 2, pegfilgrastim SC on day 3, vincristine IV on days 1 and 8, high-dose methotrexate IV over 2-4 hours on day 15, and leucovorin calcium IV beginning 24 hours after the start of methotrexate and continuing every 6 hours until level is adequate. Patients receive CNS prophylaxis of methotrexate IT, cytarabine IT, and hydrocortisone IT on day 1. Patients with high-risk disease receive an additional dose of cytarabine IT on day 3. Patients also receive G-CSF SC once daily on days 3-9. Once the methotrexate levels drops below 50 nmol/L, patients resume G-CSF SC once daily beginning on approximately day 18 and continuing until blood counts recover.
  Interventions: Biological: filgrastim; Biological: pegfilgrastim; Biological: rituximab; Drug: cyclophosphamide; Drug: cytarabine; Drug: doxorubicin hydrochloride; Drug: leucovorin calcium; Drug: liposomal cytarabine; Drug: methotrexate; Drug: therapeutic hydrocortisone; Drug: vincristine sulfate
- Regimen B (rituximab and IVAC chemotherapy) (Experimental): Patients receive rituximab IV on day 1, ifosfamide IV continuously and etoposide IV continuously over 24 hours on days 1-5, and high-dose cytarabine IV over 1-3 hours twice daily on days 1-2. Patients receive CNS prophylaxis comprising methotrexate IT and hydrocortisone IT on day 5. Patients also receive pegfilgrastim SC once 24-48 hours after completion of chemotherapy OR G-CSF SC beginning on day 6 and continuing until blood counts recover. Patients with CNS involvement (leptomeningeal and/or intraparenchymal) at diagnosis do not receive CNS prophylaxis as above. Instead, these patients receive a combination of sequential liposomal cytarabine and methotrexate IT or via an Ommaya reservoir on day 1 and then every 14 days as tolerated until completion of systemic chemotherapy.
  Interventions: Biological: filgrastim; Biological: pegfilgrastim; Biological: rituximab; Drug: cytarabine; Drug: etoposide; Drug: ifosfamide; Drug: liposomal cytarabine; Drug: methotrexate; Drug: therapeutic hydrocortisone

INTERVENTIONS:
Biological: filgrastim — given subcutaneously
Biological: pegfilgrastim — given subcutaneously
Biological: rituximab — given IV
Drug: cyclophosphamide — given IV
  Arms: Regimen A (R-CODOX-M chemotherapy)
Drug: cytarabine — given intrathecally
Drug: doxorubicin hydrochloride — given IV
  Arms: Regimen A (R-CODOX-M chemotherapy)
Drug: etoposide — given IV
  Arms: Regimen B (rituximab and IVAC chemotherapy)
Drug: ifosfamide — given IV
  Arms: Regimen B (rituximab and IVAC chemotherapy)
Drug: leucovorin calcium — given IV
  Arms: Regimen A (R-CODOX-M chemotherapy)
Drug: liposomal cytarabine — given intrathecally
Drug: methotrexate — given intrathecally
Drug: therapeutic hydrocortisone — given intrathecally
Drug: vincristine sulfate — given IV
  Arms: Regimen A (R-CODOX-M chemotherapy)

SUMMARY:
RATIONALE: Monoclonal antibodies, such as rituximab, can block cancer growth in different ways. Some block the ability of cancer cells to grow and spread. Others find cancer cells and help kill them or carry cancer-killing substances to them. Drugs used in chemotherapy work in different ways to stop the growth of cancer cells, either by killing the cells or by stopping them from dividing. Giving rituximab together with combination chemotherapy may kill more cancer cells.

PURPOSE: This phase II trial is studying how well giving rituximab together with combination chemotherapy works in treating patients with newly diagnosed, HIV-associated Burkitt's lymphoma.

DETAILED DESCRIPTION:
OBJECTIVES:

Primary

* Determine the efficacy of rituximab, cyclophosphamide, vincristine, doxorubicin hydrochloride, and high-dose methotrexate (R-CODOX-M ) alone or alternating with rituximab and ifosfamide, etoposide phosphate, and high-dose cytarabine (IVAC) and intrathecal CNS prophylaxis in patients with newly diagnosed, previously untreated, HIV-associated Burkitt's lymphoma or atypical Burkitt's lymphoma.
* Determine the safety of this regimen in these patients.

Secondary

* Evaluate downstream effectors of apoptosis as mechanisms of chemotherapy resistance and prognosis and perform exploratory analysis of their relationship to treatment effect.
* Evaluate multi-drug resistance gene expression as a mechanism of chemotherapy resistance and prognosis and perform exploratory analysis of their relationship to treatment effect.
* Confirm the use of flow cytometry in the identification of occult leptomeningeal disease and determine whether abnormal flow cytometry is predictive when CNS cytology is negative for malignant cells.
* Determine the biologic and prognostic significance of Epstein-Barr virus (EBV)-positive Burkitt's lymphoma in the highly active antiretroviral therapy era and perform exploratory analysis of their relationship to treatment effect.
* Compare genotyping in patients with HIV-associated Burkitt's lymphoma with that of patients who are HIV-negative and determine whether they are uniform in their genetic profile or whether some cases are more like diffuse large B-cell lymphoma.
* Determine if EBV detection in cerebrospinal fluid at diagnosis is predictive of leptomeningeal disease.

OUTLINE: This is a prospective, multicenter study. Patients are stratified according to risk category (low-risk vs high-risk). Patients with low-risk disease receive 3 courses of R-CODOX-M chemotherapy as described below. Patients with high-risk disease receive 4 alternating courses of R-CODOX-M/IVAC chemotherapy as described below in an A/B/A/B sequence.* Courses repeat every 21-28 days in the absence of disease progression or unacceptable toxicity.

NOTE: *In patients presenting with anasarca, pleural effusion, or ascites, methotrexate can pool causing difficulties with clearance; in this case, treatment may be given in a reverse sequence: B/A/B/A.

* Regimen A (R-CODOX-M chemotherapy): Patients receive rituximab** IV and doxorubicin hydrochloride IV over 15 minutes on day 1, cyclophosphamide IV over 30-60 minutes on days 1 and 2, pegfilgrastim subcutaneously (SC) on day 3, vincristine IV on days 1 and 8, high-dose methotrexate IV over 2-4 hours on day 15, and leucovorin calcium IV beginning 24 hours after the start of methotrexate and continuing every 6 hours until the methotrexate level is less than 50 nmol/L. Patients receive CNS prophylaxis comprising methotrexate intrathecally (IT), cytarabine IT, and hydrocortisone IT on day 1. Patients with high-risk disease receive an additional dose of cytarabine IT on day 3. Patients also receive filgrastim (G-CSF) SC once daily on days 3-9. Once the methotrexate levels drops below 50 nmol/L, patients resume G-CSF SC once daily beginning on approximately day 18 and continuing until blood counts recover.
* Regimen B (rituximab and IVAC chemotherapy): Patients receive rituximab** IV on day 1, ifosfamide IV continuously and etoposide IV continuously over 24 hours on days 1-5, and high-dose cytarabine IV over 1-3 hours twice daily on days 1-2. Patients receive CNS prophylaxis comprising methotrexate IT and hydrocortisone IT on day 5. Patients also receive pegfilgrastim SC once 24-48 hours after completion of chemotherapy OR G-CSF SC beginning on day 6 and continuing until blood counts recover.

Patients with CNS involvement (leptomeningeal and/or intraparenchymal) at diagnosis do not receive CNS prophylaxis as above. Instead, these patients receive a combination of sequential liposomal cytarabine and methotrexate IT or via an Ommaya reservoir on day 1 and then every 14 days as tolerated until completion of systemic chemotherapy.

NOTE: **Rituximab may be given up to 3 days before a chemotherapy course and anytime during the course for 3 (low-risk disease) or 4 (high-risk disease) total doses.

Patients undergo blood and cerebrospinal fluid collection and tumor biopsies periodically during study treatment for correlative studies of prognostic biomarkers predictive of survival (e.g., c-flip protein expression; p53 mutations [by immunohistochemistry (IHC)]; multidrug resistance gene expression [by IHC]; and Epstein-Barr virus in tumor DNA or cerebrospinal fluid [by polymerase chain reaction]); genotyping of Burkitt's lymphoma; and flow cytometry as a tool (by staining) for detecting occult positivity of leptomeningeal disease in Burkitt's lymphoma.

After completion of study treatment, patients are followed every 4 months for at least 2 years.

PROJECTED ACCRUAL: A total of 34 patients will be accrued for this study.

ELIGIBILITY:
DISEASE CHARACTERISTICS:

* Histologically confirmed Burkitt's lymphoma (BL) or new WHO 2009 criteria B-cell lymphoma unclassified (with features intermediated between difuse large B-cell lymphoma and BL)

  * Any stage disease
  * Newly diagnosed disease
* Meets 1 of the following criteria for disease risk:

  * Low-risk disease, defined by 1 of the following:

    * Stage I with a single focus of disease < 10 cm AND normal lactate dehydrogenase (LDH) level
    * Totally resected intra-abdominal disease only AND normal LDH post surgery
  * High-risk disease, defined as not meeting criteria for low-risk disease
* Measurable or nonmeasurable disease
* HIV-positive confirmed by enzyme-linked immunosorbent assay and Western blot OR by measurable HIV viral load
* No visceral Kaposi's sarcoma

PATIENT CHARACTERISTICS:

* Karnofsky performance status 40-100%
* Not pregnant or nursing
* Negative pregnancy test
* Fertile patients must use effective contraception
* LVEF ≥ 50% by MUGA or echocardiogram
* Creatinine ≤ 1.5 mg/dL OR creatinine clearance ≥ 60 mL/min
* Absolute neutrophil count ≥ 1,000/mm³
* Platelet count ≥ 50,000/mm³ (unless related to lymphoma)*
* Direct bilirubin ≤ 2.0 mg/dL OR total bilirubin ≤ 3.5 mg/dL AND direct bilirubin normal (if elevated bilirubin secondary to antiretroviral therapy)
* AST and ALT ≤ 3 times upper limit of normal
* No other malignancy within the past 5 years except curatively treated cutaneous basal cell or squamous cell carcinoma, carcinoma in situ of the cervix, or cutaneous Kaposi's sarcoma
* No other medical illness unrelated to non-Hodgkin's lymphoma, including any of the following:

  * Uncontrolled infection (including opportunistic infection)
  * Chronic renal insufficiency
  * Myocardial infarction within the past 6 months
  * Unstable angina
  * Cardiac arrhythmias other than chronic atrial fibrillation
* Patients with active hepatitis B infection are eligible provided they receive concurrent dual antiviral therapy NOTE: *Patients with bone marrow involvement are eligible irrespective of blood count

PRIOR CONCURRENT THERAPY:

* See Disease Characteristics
* No prior therapy for this disease except for 1 of the following :

  * Seven consecutive days of steroids alone or in combination with a non-CHOP regimen necessary for patient stabilization (e.g., cyclophosphamide and steroids steroids for normalization of disease-related hyperbilirubinemia)
  * One course of CHOP or fractionated CHOP (e.g. CODOX) with or without rituximab
* No epoetin alfa or filgrastim (G-CSF) within 24 hours of study chemotherapy
* No concurrent zidovudine

Ages: 18 Years to 120 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 34 (Actual)
Dates: Start 2006-09; Primary Completion 2011-07 (Actual); Study Completion 2013-07 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Ariela Noy, MD, Study Chair — Memorial Sloan Kettering Cancer Center; David M. Aboulafia, MD, Study Chair — Floyd & Delores Jones Cancer Institute at Virginia Mason Medical Center; Lawrence D. Kaplan, MD, Study Chair — University of California, San Francisco
Locations (13):
- United States (13):
  - Rebecca and John Moores UCSD Cancer Center, La Jolla, California
  - USC/Norris Comprehensive Cancer Center and Hospital, Los Angeles, California
  - UCLA Clinical AIDS Research and Education (CARE) Center, Los Angeles, California
  - UCSF Medical Center at Parnassus, San Francisco, California
  - Sidney Kimmel Comprehensive Cancer Center at Johns Hopkins, Baltimore, Maryland
  - Beth Israel Deaconess Medical Center, Boston, Massachusetts
  - Siteman Cancer Center at Barnes-Jewish Hospital - Saint Louis, St Louis, Missouri
  - Memorial Sloan-Kettering Cancer Center, New York, New York
  - Albert Einstein Cancer Center at Albert Einstein College of Medicine, The Bronx, New York
  - Arthur G. James Cancer Hospital and Richard J. Solove Research Institute at Ohio State University Comprehensive Cancer Center, Columbus, Ohio
  - Pennsylvania Oncology Hematology Associates, Incorporated - Philadelphia, Philadelphia, Pennsylvania
  - Floyd and Delores Jones Cancer Institute at Virginia Mason Medical Center, Seattle, Washington
  - West Virginia University Health Sciences Center - Charleston, Charleston, West Virginia

REFERENCES:
- [Result] Noy A, Lee JY, Cesarman E, Ambinder R, Baiocchi R, Reid E, Ratner L, Wagner-Johnston N, Kaplan L; AIDS Malignancy Consortium. AMC 048: modified CODOX-M/IVAC-rituximab is safe and effective for HIV-associated Burkitt lymphoma. Blood. 2015 Jul 9;126(2):160-6. doi: 10.1182/blood-2015-01-623900. Epub 2015 May 8. PMID 25957391

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Regimen A (R-CODOX-M Chemotherapy) | Regimen B (Rituximab and IVAC Chemotherapy)
Started | 2 | 32
Completed | 2 | 32
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Regimen A (R-CODOX-M Chemotherapy) | Regimen B (Rituximab and IVAC Chemotherapy) | Total
Number analyzed (Participants) | 2 | 32 | 34
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 2 | 32 | 34
  >=65 years | 0 | 0 | 0
Age, Continuous [Mean (Standard Deviation); unit: years] | 41 (8.5) | 41.4 (9.4) | 41.4 (9.2)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0 | 4 | 4
  Male | 2 | 28 | 30
Region of Enrollment [Number; unit: participants]
  United States | 2 | 32 | 34

OUTCOME MEASURES:

1. Primary Outcome: Overall Survival (OS) at 1 Year
Time Frame: 1 year post treatment
Measure: Number (95% Confidence Interval); unit: Cumulative proportion surviving at 1 yr
Arm/Group | Regimen A (R-CODOX-M Chemotherapy) | Regimen B (Rituximab and IVAC Chemotherapy)
Number analyzed (Participants) | 2 | 32
Cumulative proportion surviving at 1 yr | 1.0 [1.0 to 1.0] | 0.82 [0.62 to 0.92]

2. Secondary Outcome: Complete Response Rate
Time Frame: 6-8 weeks post treatment, every 4 months post-treatment for 2 years
Reporting Status: Not Posted

3. Secondary Outcome: Failure-free Survival (FFS)
Time Frame: 6-8 weeks post treatment, every 4 months post-treatment for 2 years
Reporting Status: Not Posted

4. Secondary Outcome: Event-free Survival (EFS)
Time Frame: 6-8 weeks post treatment, every 4 months post-treatment for 2 years
Reporting Status: Not Posted

5. Secondary Outcome: Toxicity
Time Frame: baseline through 2 years post-treatment
Reporting Status: Not Posted

6. Secondary Outcome: Incidence of Infection-related Deaths
Time Frame: baseline through 2 years post-treatment
Reporting Status: Not Posted

7. Secondary Outcome: Correlation of C-flip Expression, p53 Mutations, and Multidrug Resistance Expression With OS, FFS, and EFS
Time Frame: baseline through 2 years post-treatment
Reporting Status: Not Posted

8. Secondary Outcome: Utility of Flow Cytometry in Detecting Leptomeningeal Disease
Time Frame: baseline and 6-8 weeks post-treatment
Reporting Status: Not Posted

9. Secondary Outcome: Degree of Disconcordance Between Flow Cytometry and CNS Cytology Results
Time Frame: baseline
Reporting Status: Not Posted

10. Secondary Outcome: Biologic and Prognostic Significance of Epstein-Barr Virus (EBV) at Diagnosis and Correlation With OS, FFS, and EFS
Time Frame: baseline through 2 years post-treatment
Reporting Status: Not Posted

11. Secondary Outcome: Correlation of EBV Load Measurements With OS, FFS, and EFS
Time Frame: baseline through 2 years post-treatment
Reporting Status: Not Posted

ADVERSE EVENTS:
Arm/Group | Regimen A (R-CODOX-M Chemotherapy) | Regimen B (Rituximab and IVAC Chemotherapy)
Serious Adverse Events (participants affected / at risk) | 0/2 | 23/32
Other Adverse Events (participants affected / at risk) | 0/2 | 22/32
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Regimen A (R-CODOX-M Chemotherapy) (N=2) | Regimen B (Rituximab and IVAC Chemotherapy) (N=32)
Anemia (Blood and lymphatic system disorders) | 0 (0) | 4 (7)
Febrile neutropenia (Blood and lymphatic system disorders) | 0 (0) | 6 (8)
Acute coronary syndrome (Cardiac disorders) | 0 (0) | 1 (1)
Left ventricular systolic dysfunction (Cardiac disorders) | 0 (0) | 1 (1)
supraventricular tachycardia (Cardiac disorders) | 0 (0) | 1 (1)
Extraocular muscle paresis (Ear and labyrinth disorders) | 0 (0) | 1 (1)
Nausea (Gastrointestinal disorders) | 0 (0) | 1 (1)
Vomiting (Gastrointestinal disorders) | 0 (0) | 1 (1)
Death NOS (General disorders) | 0 (0) | 2 (2)
Fever (General disorders) | 0 (0) | 1 (1)
Catheter related infection (Infections and infestations) | 0 (0) | 1 (1)
Infections and infestations, other (Infections and infestations) | 0 (0) | 4 (5)
Lung infection (Infections and infestations) | 0 (0) | 3 (4)
Sepsis (Infections and infestations) | 0 (0) | 2 (2)
Skin infection (Infections and infestations) | 0 (0) | 1 (1)
Urinary tract infection (Infections and infestations) | 0 (0) | 1 (1)
Vascular access complication (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Cardiac tropinin I increased (Investigations) | 0 (0) | 1 (1)
Creatinine increased (Investigations) | 0 (0) | 1 (1)
Lymphocyte count decreased (Investigations) | 0 (0) | 1 (2)
Neutrophil count decreased (Investigations) | 0 (0) | 6 (11)
Platelet count decreased (Investigations) | 0 (0) | 9 (13)
White blood cell decreased (Investigations) | 0 (0) | 8 (17)
Hyperglycemia (Metabolism and nutrition disorders) | 0 (0) | 1 (2)
Tumor lysis syndrome (Metabolism and nutrition disorders) | 0 (0) | 1 (1)
Myelodysplastic syndrome (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Encephalopathy (Nervous system disorders) | 0 (0) | 1 (2)
Ischemia cerebrovascular (Nervous system disorders) | 0 (0) | 1 (1)
Transient ischemia attach (Nervous system disorders) | 0 (0) | 1 (1)
Nystagmus (Nervous system disorders) | 0 (0) | 1 (1)
Oculomotor nerve disorder (Nervous system disorders) | 0 (0) | 1 (1)
Peripheral sensory neuropathy (Nervous system disorders) | 0 (0) | 1 (1)
Acute kidney injury (Renal and urinary disorders) | 0 (0) | 1 (1)
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (2)
Pneumonitis (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Hypotension (Vascular disorders) | 0 (0) | 1 (2)
Thromboembolic event (Vascular disorders) | 0 (0) | 2 (2)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Regimen A (R-CODOX-M Chemotherapy) (N=2) | Regimen B (Rituximab and IVAC Chemotherapy) (N=32)
Anemia (Blood and lymphatic system disorders) | 0 (0) | 15 (34)
Febrile neutropenia (Blood and lymphatic system disorders) | 0 (0) | 3 (4)
Diarrhea (Gastrointestinal disorders) | 0 (0) | 2 (3)
Oral mucositis (Gastrointestinal disorders) | 0 (0) | 2 (2)
Nausea (Gastrointestinal disorders) | 0 (0) | 4 (4)
Vomiting (Gastrointestinal disorders) | 0 (0) | 5 (7)
Pain (General disorders) | 0 (0) | 3 (3)
Urinary tract infection (Infections and infestations) | 0 (0) | 2 (2)
Activated partial thromboplastin time prolonged (Investigations) | 0 (0) | 2 (2)
Alanine aminotransferase increased (Investigations) | 0 (0) | 4 (9)
Aspartate aminotransferase increased (Investigations) | 0 (0) | 6 (14)
Blood bilirubin increased (Investigations) | 0 (0) | 3 (6)
Lymphocyte count decreased (Investigations) | 0 (0) | 2 (5)
Neutrophil count decreased (Investigations) | 0 (0) | 14 (26)
Platelet count decreased (Investigations) | 0 (0) | 16 (39)
Weight loss (Investigations) | 0 (0) | 2 (2)
White blood cell count decreased (Investigations) | 0 (0) | 9 (41)
Hypercalcemia (Metabolism and nutrition disorders) | 0 (0) | 2 (2)
Hyperglycemia (Metabolism and nutrition disorders) | 0 (0) | 7 (11)
Hypocalcemia (Metabolism and nutrition disorders) | 0 (0) | 4 (8)
Hypoglycemia (Metabolism and nutrition disorders) | 0 (0) | 2 (2)
Hypokalemia (Metabolism and nutrition disorders) | 0 (0) | 8 (15)
Hyponatremia (Metabolism and nutrition disorders) | 0 (0) | 4 (9)
Hypophosphatemia (Metabolism and nutrition disorders) | 0 (0) | 5 (10)
Headache (Nervous system disorders) | 0 (0) | 4 (5)
Confusion (Psychiatric disorders) | 0 (0) | 2 (2)
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 3 (5)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2011-01-21): https://cdn.clinicaltrials.gov/large-docs/34/NCT00392834/Prot_SAP_001.pdf